CLINICAL TRIAL: NCT01976338
Title: A Randomized Double-masked, Phase III Study Assessing Ranibizumab Intravitreal Injections Versus Sham Control in Patients With Visual Impairment Due to Macular Edema (ME) Secondary to Branch Retinal Vein Occlusion (BRVO) [Blossom]
Brief Title: Ranibizumab Intravitreal Injections Versus Sham Control in Patients With Branch Retinal Vein Occlusion (BRVO)
Acronym: Blossom
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002E2303
Record Dates: First submitted 2013-10-18; First posted 2013-11-05 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Macular Edema Secondary to Branch Retinal Vein Occlusion
Keywords: BRVO; macular edema; vision impairment; retinal vein occlusion; ranibizumab; branch retinal vein occlusion; anti-VEGF therapy; RFB002
MeSH Terms: conditions — Macular Edema; Vision Disorders; Retinal Vein Occlusion | interventions — Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab 0.5 mg (Experimental): PRN Intravitreal injection
  Interventions: Drug: Ranibizumab 0.5 mg
- Sham injection (Sham Comparator): As of Month 6 ranibizumab 0.5 mg PRN intravitreal injection
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: Ranibizumab 0.5 mg — intravitreal injection of 0.05 ml
  Arms: Ranibizumab 0.5 mg
Other: Sham injection — Sham intravitreal injection
  Other Names: Sham
  Arms: Sham injection

SUMMARY:
Provided efficacy and safety data on intravitreal injections of ranibizumab 0.5 mg in patients with visual impairment due to macular edema secondary to BRVO

ELIGIBILITY:
Inclusion Criteria:

• Patients with visual impairment secondary to branch retinal vein occlusion (BRVO) with a BCVA between 19 and 73 letters in one eye and at least 35 letters in the other eye.

Exclusion Criteria:

* Pregnant or nursing women or women of child bearing potential without unless using an effective contraception
* Stroke or myocard infarction within 3 months prior to study
* History of malignancy within the past 5 years
* Uncontrolled hypertension
* Active infection or inflammation in any eye
* use of corticosteroids for at least 30 days in the last 6 months
* treatment with anti-angiogenic drugs in any eye within last 3 months
* Panretinal or focal/drid laser photocoagulation within the last few months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2016-03-28 (Actual); Study Completion 2016-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- China (17):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nantong, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- Indonesia (2):
  - Novartis Investigative Site, Jakarta, Jakarta Special Capital Region
  - Novartis Investigative Site, Bandung, West Java
- Philippines (2):
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, San Juan City, Philippines
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Taipei
- Vietnam (2):
  - Novartis Investigative Site, Hanoi, Vietnam
  - Novartis Investigative Site, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Wei W, Weisberger A, Zhu L, Cheng Y, Liu C; BLOSSOM Study Group. Efficacy and Safety of Ranibizumab in Asian Patients with Branch Retinal Vein Occlusion: Results from the Randomized BLOSSOM Study. Ophthalmol Retina. 2020 Jan;4(1):57-66. doi: 10.1016/j.oret.2019.08.001. Epub 2019 Aug 13. PMID 31902472

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of the following three periods (Screening period: Day -14 to Day -1; treatment period: Day 1 to Month 11; post-treatment Follow-Up period: Month 11 to Month 12). At Baseline (Visit 2, Day 1), eligible patients were randomized in a 2:1 ratio into respective treatment arms
Period: Overall Study
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Started | 190 | 93
Completed 6 Months | 185 | 91
Discontinued Study Prior to 6 Months | 5 | 2
Completed | 177 (12 months) | 89 (12 months)
Not Completed | 13 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Adverse Event | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg | Sham Injection | Total
Number analyzed (Participants) | 190 | 93 | 283
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (10.14) | 56.8 (10.03) | 56.9 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 38 | 139
  Male | 89 | 55 | 144

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Best Corrected Visual Acuity (BCVA) From Baseline to Month 1 Through Month 6
Description: Best Corrected Visual Acuity (BCVA) was assessed in a sitting position using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters. Mean Visual Acuity was averaged over all monthly assessments from month 1 to month 6 and compared to Baseline.
Time Frame: Baseline to Month 1 through Month 6
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment group they had been assigned to at randomization. Mean value interpolation and last observation carried forward (MV-LOCF)
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 189 | 93
Letters | 12.5 (8.34) | 5.0 (9.18)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Sham Injection; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Average Change of Best Corrected Visual Acuity (BCVA) in Patients From Baseline to Month 1 Through Month 12
Description: Best Corrected Visual Acuity (BCVA) was assessed in a sitting position using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters. Mean Visual Acuity was averaged over all monthly assessments from month 1 to month 12 and compared to Baseline
Time Frame: Baseline to Month 1 through Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 189 | 93
Letters | 14.0 (8.99) | 7.7 (9.41)

3. Secondary Outcome: Best Corrected Visual Acuity (BCVA) Change Over Time
Description: as for outcome 2
Time Frame: Month 1 through Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 189 | 93
Letters
  Month 1 | 9.5 (8.26) | 1.7 (8.70)
  Month 2 | 11.7 (8.39) | 3.7 (8.81)
  Month 3 | 12.9 (8.81) | 5.1 (10.10)
  Month 4 | 13.4 (9.72) | 6.0 (10.44)
  Month 5 | 13.6 (10.24) | 6.5 (11.53)
  Month 6 | 14.0 (10.75) | 7.0 (12.75)
  Month 7 | 14.7 (10.62) | 8.5 (10.97)
  Month 8 | 14.9 (10.52) | 10.4 (10.97)
  Month 9 | 14.8 (10.43) | 10.3 (10.78)
  Month 10 | 15.8 (10.67) | 11.2 (11.12)
  Month 11 | 15.8 (10.42) | 11.1 (10.48)
  Month 12 | 16.4 (10.95) | 11.3 (11.11)

4. Secondary Outcome: Number of Participants With a Best Corrected Visual Acuity (BCVA) Improvement of ≥5, ≥10, ≥15, and ≥30 Letters Over Time
Description: Best Corrected Visual Acuity (BCVA) was assessed in a sitting position using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters
Time Frame: Baseline to month 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 190 | 93
Participants
  Month 1 Gain of >=5 letters | 139 | 33
  Month 1 Gain of >=10 letters | 86 | 12
  Month 1 Gain of >=15 letters | 43 | 3
  Month 1 Gain of >=30 letters | 2 | 0
  Month 2 Gain of >=5 letters | 156 | 44
  Month 2 Gain of >=10 letters | 113 | 21
  Month 2 Gain of >=15 letters | 72 | 6
  Month 2 Gain of >=30 letters | 6 | 2
  Month 3 Gain of >=5 letters | 162 | 49
  Month 3 Gain of >=10 letters | 116 | 29
  Month 3 Gain of >=15 letters | 76 | 16
  Month 3 Gain of >=30 letters | 8 | 0
  Month 4 Gain of >=5 letters | 159 | 55
  Month 4 Gain of >=10 letters | 122 | 32
  Month 4 Gain of >=15 letters | 83 | 16
  Month 4 Gain of >=30 letters | 11 | 2
  Month 5 Gain of >=5 letters | 159 | 60
  Month 5 Gain of >=10 letters | 127 | 40
  Month 5 Gain of >=15 letters | 83 | 19
  Month 5 Gain of >=30 letters | 15 | 2
  Month 6 Gain of >=5 letters | 163 | 58
  Month 6 Gain of >=10 letters | 129 | 47
  Month 6 Gain of >=15 letters | 88 | 25
  Month 6 Gain of >=30 letters | 16 | 3
  Month 7 Gain of >=5 letters | 162 | 63
  Month 7 Gain of >=10 letters | 135 | 49
  Month 7 Gain of >=15 letters | 93 | 28
  Month 7 Gain of >=30 letters | 16 | 3
  Month 8 Gain of >=5 letters | 168 | 66
  Month 8 Gain of >=150 letters | 130 | 52
  Month 8 Gain of >=15 letters | 94 | 33
  Month 8 Gain of >=30 letters | 17 | 4
  Month 9 Gain of >=5 letters | 163 | 67
  Month 9 Gain of >=10 letters | 139 | 52
  Month 9 Gain of >=15 letters | 90 | 32
  Month 9 Gain of >=30 letters | 17 | 4
  Month 10 Gain of >=5 letters | 169 | 68
  Month 10 Gain of >=10 letters | 143 | 53
  Month 10 Gain of >=15 letters | 97 | 37
  Month 10 Gain of >=30 letters | 22 | 7
  Month 11 Gain of >=5 letters | 172 | 67
  Month 11 Gain of >=10 letters | 141 | 56
  Month 11 Gain of >=15 letters | 103 | 36
  Month 11 Gain of >=30 letters | 19 | 4
  Month 12 Gain of >=5 letters | 171 | 72
  Month 12 Gain of >=10 letters | 142 | 56
  Month 12 Gain of >=15 letters | 105 | 36
  Month 12 Gain of >=30 letters | 24 | 5

5. Secondary Outcome: Number of Participants With Best Corrected Visual Acuity (BCVA)Loss of 15 Letters in the Study Eye
Description: Visual acuity (VA) was assessed at every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. This outcome measure describes for each post-baseline month whether or not a patient lost less than 15 letters of VA as compared with baseline.
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 190 | 93
Participants
  Month 1, Loss of < 15 letters | 188 | 89
  Month 2, Loss of < 15 letters | 189 | 90
  Month 3, Loss of < 15 letters | 189 | 88
  Month 4, Loss of < 15 letters | 189 | 88
  Month 5, Loss of < 15 letters | 189 | 88
  Month 6, Loss of < 15 letters | 188 | 89
  Month 7, Loss of < 15 letters | 188 | 91
  Month 8, Loss of < 15 letters | 188 | 92
  Month 9, Loss of < 15 letters | 187 | 93
  Month 10, Loss of < 15 letters | 188 | 92
  Month 11, Loss of < 15 letters | 187 | 93
  Month 12, Loss of < 15 letters | 187 | 91

6. Secondary Outcome: Change in Central-Sub-Field- Thickness (CSFT) Over Time
Description: OCT (optical coherence tomography) was used to assess CSFT (Central Sub-Field Thickness) representing the average retinal thickness of the circular area within 1 mm diameter around the foveal center
Time Frame: Month 1 to month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 188 | 93
µm
  Month 1 | -261.1 (171.95) | -42.4 (171.88)
  Month 2 | -274.8 (174.17) | -93.1 (187.14)
  Month 3 | -282.2 (175.86) | -155.3 (209.37)
  Month 4 | -254.7 (183.87) | -193.2 (221.58)
  Month 5 | -258.6 (180.57) | -203.2 (218.02)
  Month 6 | -264.1 (168.64) | -206.6 (221.85)
  Month 7 | -265.4 (179.06) | -289.8 (228.03)
  Month 8 | -263.8 (179.38) | -286.1 (236.75)
  Month 9 | -266.7 (182.60) | -287.9 (237.61)
  Month 10 | -268.4 (173.71) | -282.9 (239.98)
  Month 11 | -270.6 (184.34) | -290.3 (227.47)
  Month 12 | -273.4 (184.33) | -282.9 (233.69)

7. Secondary Outcome: Change in Total Area of Fluorescein Leakage (Center Subfield) From Baseline Over Time
Description: Fluorescein leakage area was assessed using Fluorescein angiography (FA) in conjunction with 7-field color fundus photography (CF) at Screening, Month 3, Month 6 and End of Study visit for both eyes
Time Frame: month 3, 6 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 186 | 90
mm^2
  Month 3 | -0.400 (0.3576) | -0.026 (0.3387)
  Month 6 | -0.356 (0.3983) | -0.055 (0.4060)
  Month 12 | -0.391 (0.3716) | -.0208 (0.4075)

8. Secondary Outcome: Change in Total Area of Fluorescein Leakage (Inner Subfield) From Baseline Over Time
Description: as for outcome 7
Time Frame: Months 3, 6 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 186 | 90
mm^2
  Month 3 | -1.869 (1.8071) | 0.111 (1.5497)
  Month 6 | -1.642 (1.9570) | -0.078 (1.6856)
  Month 12 | -1.732 (1.8059) | -0.823 (1.9650)

9. Secondary Outcome: Change in Total Area of Fluorescein Leakage (Outer Subfield) From Baseline Over Time
Description: as for outcome 7
Time Frame: Months 3, 6 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 186 | 90
mm^2
  Month 3 | -4.994 (5.4066) | -0.600 (3.6646)
  Month 6 | -4.654 (5.7504) | -0.836 (4.2819)
  Month 12 | -5.078 (5.9568) | -2.797 (5.3702)

10. Secondary Outcome: Change From Baseline in NEI-VFQ-25 Composite and Subscale Scores at Month 3, Month 6 and Month 12
Description: The VFQ-25 consists of 25 vision related questions across 11 vision related subscales, including general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision and peripheral vision, and a general health rating. Items are converted to a 0-100 scale on each subscale and for the composite score where higher scores represents better functioning.
Time Frame: Baseline, months 3, 6 and 12
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment group they had been assigned to at randomization. n=the number of patients with a value for both baseline and the specific post-baseline visit.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Ranibizumab 0.5 mg | Sham Injection
Number analyzed (Participants) | 190 | 93
Scores on a Scale
  Change from Baseline at M3 (n=187,91) | 5.8 (10.85) | -1.1 (11.21)
  Change from Baseline at M6 (n=185,88) | 7.7 (11.88) | 0.1 (13.95)
  Change from Baseline at M12 (n=176,88) | 9.6 (13.45) | 3.3 (13.52)

ADVERSE EVENTS:
Description: The Safety Set consisted of all patients who received at least one application of study treatment and had at least one post-Baseline safety assessment. Patients were analyzed according to the treatment received. The statement that a patient had no AEs also constituted a safety assessment.
Groups:
- Sham With Ranibizumab 0.5 mg: As of Month 6 ranibizumab 0.5 mg PRN intravitreal injection
- Sham Without Ranibizumab 0.5 mg: sham + ranibizumab 0.5 mg PRN as of Month 6 (hereafter referred to as sham group up to Month 6 and sham with ranibizumab or sham without ranibizumab after Month 6)
Arm/Group | Ranibizumab 0.5 mg | Sham With Ranibizumab 0.5 mg | Sham Without Ranibizumab 0.5 mg
Serious Adverse Events (participants affected / at risk) | 13/190 | 3/66 | 3/26
Other Adverse Events (participants affected / at risk) | 119/190 | 46/66 | 14/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=190) | Sham With Ranibizumab 0.5 mg (N=66) | Sham Without Ranibizumab 0.5 mg (N=26)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Macular hole (Eye disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cluster headache (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 2 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=190) | Sham With Ranibizumab 0.5 mg (N=66) | Sham Without Ranibizumab 0.5 mg (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1 | 0
Coronary artery disease (Cardiac disorders) | 4 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 1 | 0
Conjunctival deposit (Eye disorders) | 2 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 20 | 4 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Corneal epithelium defect (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 3 | 0 | 1
Eye irritation (Eye disorders) | 1 | 2 | 0
Eye pain (Eye disorders) | 10 | 1 | 0
Eye pruritus (Eye disorders) | 4 | 1 | 0
Eye swelling (Eye disorders) | 2 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 1 | 1
Foreign body sensation in eyes (Eye disorders) | 6 | 1 | 1
Glare (Eye disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 3 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 2 | 0
Macular fibrosis (Eye disorders) | 6 | 1 | 0
Ocular hyperaemia (Eye disorders) | 2 | 0 | 0
Ocular hypertension (Eye disorders) | 3 | 0 | 0
Open angle glaucoma (Eye disorders) | 2 | 0 | 0
Retinal fibrosis (Eye disorders) | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 3 | 3 | 0
Retinal ischaemia (Eye disorders) | 7 | 3 | 1
Retinal neovascularisation (Eye disorders) | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 1 | 0
Vision blurred (Eye disorders) | 3 | 2 | 0
Visual acuity reduced (Eye disorders) | 1 | 2 | 0
Vitreous detachment (Eye disorders) | 3 | 1 | 0
Vitreous floaters (Eye disorders) | 4 | 2 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Vitreous opacities (Eye disorders) | 3 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 3 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 6 | 2 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0 | 0
Conjunctivitis (Infections and infestations) | 5 | 1 | 1
Gingivitis (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 23 | 8 | 3
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 2 | 1 | 0
Blood pressure increased (Investigations) | 3 | 0 | 0
Glucose urine present (Investigations) | 0 | 0 | 1
Haemoglobin urine present (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 10 | 1 | 0
Optic nerve cup/disc ratio increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 1 | 0
Visual acuity tests abnormal (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 6 | 2 | 0
Headache (Nervous system disorders) | 11 | 2 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 16 | 8 | 4

LIMITATIONS AND CAVEATS:
One patient was randomized to the ranibizumab group but received no study treatment during the study period and discontinued the study after Visit 2. Therefore, excluded from the Safety set

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety